CLINICAL TRIAL: NCT04208789
Title: Artificial Neural Network as Diagnostic Tools For Rifampicin-Resistant Tuberculosis In Indonesia: A Predictive Model Study and Economic Evaluation
Brief Title: Artificial Inteligent for Diagnosing Drug-Resistant Tuberculosis
Status: Completed | Type: Observational
Sponsor: Hasanuddin University (Other)
Collaborators: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Bumi Herman, Researcher, Hasanuddin University
Other Study IDs: 0111190912
Record Dates: First submitted 2019-12-06; First posted 2019-12-23 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: MDR Tuberculosis; Resistance to Tuberculostatic Drugs
Keywords: Artificial Neural Network; GeneXpert MTB/RIF; Drug-Resistant Tb; Diagnosis
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive Rifampicin-Resistant Tuberculosis: All suspected cases that yielded Positive Rifampicin-Resistant Tuberculosis under the Gold-Standard Test (Culture on Lowenstein-Jensen Medium)
  Interventions: Diagnostic Test: Rapid Molecular Drug-Resistant Tuberculosis Test; Other: Artificial Intelligent Model; Diagnostic Test: Drug Susceptibility Test
- Negative Rifampicin-Resistant Tuberculosis: All suspected cases that yielded Negative Rifampicin-Resistant Tuberculosis under the Gold-Standard Test (Culture on Lowenstein-Jensen Medium)
  Interventions: Diagnostic Test: Rapid Molecular Drug-Resistant Tuberculosis Test; Other: Artificial Intelligent Model; Diagnostic Test: Drug Susceptibility Test

INTERVENTIONS:
Diagnostic Test: Rapid Molecular Drug-Resistant Tuberculosis Test — GeneXpert MTB/RIF assay is a nucleic acid amplification (NAA) test which simultaneously detects DNA of Mycobacterium tuberculosis complex (MTBC) and resistance to rifampin (RIF) (i.e. mutation of the rpoB gene) in less than two hours. This system integrates and automates sample processing, nucleic acid amplification, and detection of the target sequences. The primers in the XpertMTB/RIF assay amplify a portion of the rpoB gene containing the 81 base pair "core" region. The probes are able to differentiate between the conserved wild-type sequence and mutations in the core region that is associated with rifampicin resistance. The output of this procedure is detected, undetected, or indeterminate.
  Other Names: GeneXpert MTB/RIF
Other: Artificial Intelligent Model — The artificial intelligent model is a model that developed from several associated factors with machine learning and deep learning method in order to classify the possibility of drug-resistant tuberculosis. The Artificial neural network will be built using deep learning software.
  Other Names: Artificial Neural Network
Diagnostic Test: Drug Susceptibility Test — This procedure uses Löwenstein-Jensen (LJ) medium to determine whether the isolates of M. tuberculosis are susceptible to anti-TB agents. Media containing the critical concentration of the anti-TB agent is inoculated with a dilution of a culture suspension (usually a 10-2 dilution of a MacFarland 1 suspension) and control media without the anti-TB agent is inoculated with usually a 10-4 dilution of a MacFarland 1 suspension. Growth (i.e. a number of colonies) on the agent-containing media is compared to the growth on the agent-free control media. The ratio of the number of colonies on the medium containing the anti-TB agent to the number of colonies (corrected for the dilution factor) on the medium without the anti-TB agent is calculated, and the proportion is expressed as a percentage. Provisional results for susceptible isolates may be read after 3-4 weeks of incubation; definitive results may be read after 6 weeks of incubation. Resistance may be reported within 3-4 weeks.
  Other Names: Lowenstein-Jensen Medium Drug Susceptibility Test

SUMMARY:
Title: Artificial Neural Network as Diagnostic Tools For Rifampicin-Resistant Tuberculosis In Indonesia. A Predictive Model Study and Economic Evaluation.

Background: Drug-resistant tuberculosis has become a global threat particularly in Indonesia. The need to increase detection, followed by appropriate treatment is a concern in dealing with these cases. The rapid molecular test (specifically for detecting rifampicin-resistant) is now being utilized in health care service, particularly at primary care level with some challenges including the lack of quality control (including how to obtained and treat the specimen properly prior to the examination) which then, affect the reliability of the results. Drug-Susceptibility Test (DST) is still, the gold standard in diagnosing drug-resistant tuberculosis but this procedure is time-consuming and costly. The artificial intelligent including data exploration and modeling is a promising method to classify potential drug-resistant cases based on the association of several factors.

Objective :

1. To develop a model using an artificial intelligence approach that is able to classify the possibility of rifampicin-resistant tuberculosis.
2. To assess the diagnostic ability and the accuracy of the model in comparison to existing rapid test and the gold standard
3. To evaluate the cost-effectiveness evaluation of Artificial Neural Network model in Web-Based Application in comparison with the standard diagnostic tools

Methodology

1. A cross-sectional study involving all suspected drug-resistant tuberculosis cases that being referred to the study center to undergo rapid molecular test and DST test over the past 5 years.
2. A comprehensive, retrospective medical records assessment and tuberculosis individual report will be performed to obtain a variable of interest.
3. Questionnaire assessment for confirmation of insufficient information.
4. Model Building through machine learning and deep learning procedure
5. Model Validation and testing using training data set and data from the different study center

Hypothesis :

Artificial Intelligent Model will yield a similar or superior result of diagnostic ability compare the Rapid Molecular Test according to the Drug-Susceptibility Test. (Superiority Trial)

DETAILED DESCRIPTION:
PROCEDURE

1. Under the permission granted by the study centers, the team will obtain the medical records of all eligible cases within the past 5 years
2. The investigators then collect the information of interest variable/parameter which obtained by history taking and further examinations and also medical Billing and Hospital pay per service. For participants with Health Insurance, the direct spending for treatment will be based on INA-CBGs (case-based group) payment. This data then will be recorded in an electronic database.

   Parameter for model development :

   Host-based :
   1. Presence of Diabetes Mellitus (Including years of being diagnosed, HbA1c Before DST examination and treatment, medication either insulin or oral anti-diabetic)
   2. Presence of HIV ((Including years of being diagnosed, CD4 level Before DST examination and treatment, and anti-retroviral medication)
   3. Tobacco cessation (Brinkman Index)
   4. Alcohol consumption
   5. History of Immunosuppressant use (steroid)
   6. Presence of other diseases (cancer, stroke, cardiovascular disease)
   7. History of drug abuse
   8. History of adverse drug reaction during tuberculosis treatment
   9. Adherence of previous tuberculosis therapy
   10. Presence of COPD
   11. Body Mass Index

   Environment
   1. History of Contact with Tuberculosis Patients
   2. Healthy Index of Living Environment (Household crowds)

   Agent
   1. Level of Bacterial Smear Before DST
   2. Extension of Lesion in Chest X-Ray
   3. Presence of Cavitation

   Sociodemographic Factors
   1. Age
   2. Gender
   3. Education
   4. Income Level
   5. Health Insurance
   6. Marital Status
   7. Employment Status
3. For incomplete information, a confirmation to the health center that was referring the cases will be done using the Tuberculosis Registration or questionnaire.
4. The model building will be done using an Artificial Intelligent Model in R. A selected model is an Artificial Neural Network either using Radial Base Function or multi-layer perceptron. Several important procedures including :

   1. Determine Significant Parameter
   2. Dealing with Insufficient and Imbalanced data class (over or under-sampling)
   3. Normalization (Batch, Min-Max)
   4. Layer and design
   5. Training and test distribution (70:30)
   6. Model Selection
5. External Validation will be done to the appointed study center. Precision: (true positive + True Negative)/All cases
6. The Incremental Cost-Effectiveness Ratio Simulation will be done, comparing the best model versus the gold standard and GeneXpert yielding a saving per unit of effectiveness

ELIGIBILITY:
Inclusion criteria:

1. Default cases under WHO criteria
2. Failure cases under WHO criteria
3. Physician-referred cases for presumptive drug-resistant TB as follows :

With or without immunocompromised condition, With or without any adverse reaction of anti TB drug, With or without any comorbidities (such as diabetes mellitus, heart disease)

Exclusion Criteria:

1. Incomplete Information on Rapid Molecular Test Results, and Culture Results
2. Participants or family are unable/unwilling to provide additional information obtained through questionnaire

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All suspected/presumptive Drug-Resistant Tuberculosis cases that were sent to the appointed Study Center within the last 3 years
Sampling Method: Non-Probability Sample
Enrollment: 524 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-02 (Actual)

PRIMARY OUTCOMES:
Accuracy of Artificial Intelligent Model to Drug Susceptibility Test Results | through study completion, an average of 1 year
  The accuracy is the number of correct cases (the results obtained by the model is the same as obtained by culture) predicted by the model per total cases.

SECONDARY OUTCOMES:
Accuracy of Rapid Molecular Drug Resistant Tuberculosis test to Drug Susceptibility Test Results | through study completion, an average of 1 year
  The accuracy is the number of correct cases (the results obtained by the GeneXpert MTB/RIF is the same as obtained by culture) predicted by the model per total cases.

OTHER OUTCOMES:
Diagnostic Ability of Artificial Intelligent Model to Drug Susceptibility Test Results | through study completion, an average of 1 year
  Sensitivity, Specificity, Negative Predictive Value and Positive Predictive value of Artificial Intelligent Model to Drug Susceptibility Test Results

CONTACTS AND LOCATIONS:
Overall Officials: Sathirakorn Pongpanich, Prof, Study Director — Chulalongkorn University; Wandee Sirichokchatchawan, Ph.D, Principal Investigator — Chulalongkorn University; Bumi Herman, MD, Principal Investigator — Hasanuddin University
Locations (5):
- Indonesia (5):
  - Kanudjoso Djatiwibowo General Hospital, Balikpapan, East Kalimantan
  - Tarakan General Hospital, Tarakan, North Kalimantan
  - Wahidin Sudirohusodo General Hospital, Makassar, South Sulawesi
  - Labuang Baji General Hospital, Makassar, South Sulawesi
  - Balai Besar Kesehatan Paru Masyarakat, Makassar, South Sulawesi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] GBD Tuberculosis Collaborators. The global burden of tuberculosis: results from the Global Burden of Disease Study 2015. Lancet Infect Dis. 2018 Mar;18(3):261-284. doi: 10.1016/S1473-3099(17)30703-X. Epub 2017 Dec 7. PMID 29223583
- [Background] Dean AS, Cox H, Zignol M. Epidemiology of Drug-Resistant Tuberculosis. Adv Exp Med Biol. 2017;1019:209-220. doi: 10.1007/978-3-319-64371-7_11. PMID 29116637
- [Background] Kendall EA, Azman AS, Cobelens FG, Dowdy DW. MDR-TB treatment as prevention: The projected population-level impact of expanded treatment for multidrug-resistant tuberculosis. PLoS One. 2017 Mar 8;12(3):e0172748. doi: 10.1371/journal.pone.0172748. eCollection 2017. PMID 28273116
- [Background] Dheda K, Gumbo T, Maartens G, Dooley KE, McNerney R, Murray M, Furin J, Nardell EA, London L, Lessem E, Theron G, van Helden P, Niemann S, Merker M, Dowdy D, Van Rie A, Siu GK, Pasipanodya JG, Rodrigues C, Clark TG, Sirgel FA, Esmail A, Lin HH, Atre SR, Schaaf HS, Chang KC, Lange C, Nahid P, Udwadia ZF, Horsburgh CR Jr, Churchyard GJ, Menzies D, Hesseling AC, Nuermberger E, McIlleron H, Fennelly KP, Goemaere E, Jaramillo E, Low M, Jara CM, Padayatchi N, Warren RM. The epidemiology, pathogenesis, transmission, diagnosis, and management of multidrug-resistant, extensively drug-resistant, and incurable tuberculosis. Lancet Respir Med. 2017 Mar 15:S2213-2600(17)30079-6. doi: 10.1016/S2213-2600(17)30079-6. Online ahead of print. PMID 28344011
- [Background] Collins D, Hafidz F, Mustikawati D. The economic burden of tuberculosis in Indonesia. Int J Tuberc Lung Dis. 2017 Sep 1;21(9):1041-1048. doi: 10.5588/ijtld.16.0898. PMID 28826455
- [Background] Falzon D, Mirzayev F, Wares F, Baena IG, Zignol M, Linh N, Weyer K, Jaramillo E, Floyd K, Raviglione M. Multidrug-resistant tuberculosis around the world: what progress has been made? Eur Respir J. 2015 Jan;45(1):150-60. doi: 10.1183/09031936.00101814. Epub 2014 Sep 26. PMID 25261327
- [Background] Falzon D, Jaramillo E, Wares F, Zignol M, Floyd K, Raviglione MC. Universal access to care for multidrug-resistant tuberculosis: an analysis of surveillance data. Lancet Infect Dis. 2013 Aug;13(8):690-7. doi: 10.1016/S1473-3099(13)70130-0. Epub 2013 Jun 4. PMID 23743044
- [Background] van Kampen SC, Susanto NH, Simon S, Astiti SD, Chandra R, Burhan E, Farid MN, Chittenden K, Mustikawati DE, Alisjahbana B. Effects of Introducing Xpert MTB/RIF on Diagnosis and Treatment of Drug-Resistant Tuberculosis Patients in Indonesia: A Pre-Post Intervention Study. PLoS One. 2015 Jun 15;10(6):e0123536. doi: 10.1371/journal.pone.0123536. eCollection 2015. PMID 26075722
- [Background] Soeroto AY, Lestari BW, Santoso P, Chaidir L, Andriyoko B, Alisjahbana B, van Crevel R, Hill PC. Evaluation of Xpert MTB-RIF guided diagnosis and treatment of rifampicin-resistant tuberculosis in Indonesia: A retrospective cohort study. PLoS One. 2019 Feb 28;14(2):e0213017. doi: 10.1371/journal.pone.0213017. eCollection 2019. PMID 30818352
- [Background] Prada-Medina CA, Fukutani KF, Pavan Kumar N, Gil-Santana L, Babu S, Lichtenstein F, West K, Sivakumar S, Menon PA, Viswanathan V, Andrade BB, Nakaya HI, Kornfeld H. Systems Immunology of Diabetes-Tuberculosis Comorbidity Reveals Signatures of Disease Complications. Sci Rep. 2017 May 17;7(1):1999. doi: 10.1038/s41598-017-01767-4. PMID 28515464
- [Background] Pradipta IS, Forsman LD, Bruchfeld J, Hak E, Alffenaar JW. Risk factors of multidrug-resistant tuberculosis: A global systematic review and meta-analysis. J Infect. 2018 Dec;77(6):469-478. doi: 10.1016/j.jinf.2018.10.004. Epub 2018 Oct 16. PMID 30339803
- [Background] Wang MG, Huang WW, Wang Y, Zhang YX, Zhang MM, Wu SQ, Sandford AJ, He JQ. Association between tobacco smoking and drug-resistant tuberculosis. Infect Drug Resist. 2018 Jun 12;11:873-887. doi: 10.2147/IDR.S164596. eCollection 2018. PMID 29928135
- [Background] Alipanah N, Jarlsberg L, Miller C, Linh NN, Falzon D, Jaramillo E, Nahid P. Adherence interventions and outcomes of tuberculosis treatment: A systematic review and meta-analysis of trials and observational studies. PLoS Med. 2018 Jul 3;15(7):e1002595. doi: 10.1371/journal.pmed.1002595. eCollection 2018 Jul. PMID 29969463
- [Background] Tegegne BS, Mengesha MM, Teferra AA, Awoke MA, Habtewold TD. Association between diabetes mellitus and multi-drug-resistant tuberculosis: evidence from a systematic review and meta-analysis. Syst Rev. 2018 Oct 15;7(1):161. doi: 10.1186/s13643-018-0828-0. PMID 30322409
- [Background] Darsey JA, Griffin WO, Joginipelli S, Melapu VK. Architecture and biological applications of artificial neural networks: a tuberculosis perspective. Methods Mol Biol. 2015;1260:269-83. doi: 10.1007/978-1-4939-2239-0_17. PMID 25502388
- [Background] Souza Filho JBOE, Sanchez M, Seixas JM, Maidantchik C, Galliez R, Moreira ADSR, da Costa PA, Oliveira MM, Harries AD, Kritski AL. Screening for active pulmonary tuberculosis: Development and applicability of artificial neural network models. Tuberculosis (Edinb). 2018 Jul;111:94-101. doi: 10.1016/j.tube.2018.05.012. Epub 2018 May 19. PMID 30029922
- [Background] Dande P, Samant P. Acquaintance to Artificial Neural Networks and use of artificial intelligence as a diagnostic tool for tuberculosis: A review. Tuberculosis (Edinb). 2018 Jan;108:1-9. doi: 10.1016/j.tube.2017.09.006. Epub 2017 Sep 20. PMID 29523307
- [Background] de O Souza Filho JB, de Seixas JM, Galliez R, de Braganca Pereira B, de Q Mello FC, Dos Santos AM, Kritski AL. A screening system for smear-negative pulmonary tuberculosis using artificial neural networks. Int J Infect Dis. 2016 Aug;49:33-9. doi: 10.1016/j.ijid.2016.05.019. Epub 2016 May 24. PMID 27235086
- [Derived] Herman B, Sirichokchatchawan W, Pongpanich S, Nantasenamat C. Development and performance of CUHAS-ROBUST application for pulmonary rifampicin-resistance tuberculosis screening in Indonesia. PLoS One. 2021 Mar 25;16(3):e0249243. doi: 10.1371/journal.pone.0249243. eCollection 2021. PMID 33765092